CLINICAL TRIAL: NCT07165977
Title: The Impact of an Anti-inflammatory Probiotic Supplementation on Cognitive Functioning in the Elderly Population - the Moderating Role of the Dietary Patterns and Gut Microbiota
Brief Title: Anti-inflammatory Probiotics in Cognitive Functioning
Acronym: CoProM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Sanprobi Sp. z o. o. (Unknown); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Aneta Brzezicka, Associate professor, Head of the Neurocognitive Research Center at SWPS University, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Cognition-Probiotic-Microbiota; 2021/43/O/HS6/02074 (Other Grant/Funding Number: National Science Centre Poland)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Memory Decline; Cognitive Decline; Cognitive Aging
Keywords: dietary patterns; probiotic intervention; cognitive functioning; EEG; ERP; gut microbiota; gut brain axis
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, and placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anti-inflammatory diet + probiotic first (Experimental): This is a group of participants whose everyday dietary pattern was assessed as anti-inflammatory based on the Shivappa et al. (2014) equation, and who will receive probiotics during the first 3 months of the study.
  Interventions: Dietary Supplement: Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52) then placebo
- Anti-inflammatory diet + placebo first (Experimental): This is a group of participants whose everyday dietary pattern was assessed as anti-inflammatory based on the Shivappa et al. (2014) equation, and who will receive placebo during the first 3 months of the study.
  Interventions: Dietary Supplement: Placebo Supplementation then Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52)
- Pro-inflammatory diet + probiotic first (Experimental): This is a group of participants whose everyday dietary pattern was assessed as pro-inflammatory based on the Shivappa et al. (2014) equation, and who will receive probiotics during the first 3 months of the study.
  Interventions: Dietary Supplement: Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52) then placebo
- Pro-inflammatory diet + placebo first (Experimental): This is a group of participants whose everyday dietary pattern was assessed as pro-inflammatory based on the Shivappa et al. (2014) equation, and who will receive placebo during the first 3 months of the study.
  Interventions: Dietary Supplement: Placebo Supplementation then Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52)

INTERVENTIONS:
Dietary Supplement: Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52) then placebo — Each participant will take a probiotic mixture containing Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52 and excipients: potato starch, magnesium stearate, and the capsule shell of hydroxypropyl methylcellulose. (Sanprobi Stress; Sanprobi sp. z o.o., sp.k., Szczecin, Poland) for 3 months.
  * Dosage: One capsule per day, containing 3 × 10⁹ (3 billion) CFU*.
  * Instructions: Take before 1:00 PM. Do not consume hot drinks immediately after taking the capsule.
  After completion of the first phase, each participant will take a probiotic containing only the excipients, i.e. maize starch, maltodextrins, and the capsule shell for another 3 months.
  * Dosage: One capsule per day.
  * Instructions: Take before 1:00 PM. Do not consume hot drinks immediately after taking the capsule.
  * CFU = Colony Forming Units
  Arms: Anti-inflammatory diet + probiotic first; Pro-inflammatory diet + probiotic first
Dietary Supplement: Placebo Supplementation then Probiotic Supplementation (Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52) — Each participant will take a probiotic containing only the excipients, i.e. maize starch, maltodextrins, and the capsule shell for 3 months.
  * Dosage: One capsule per day.
  * Instructions: Take before 1:00 PM. Do not consume hot drinks immediately after taking the capsule.
  After completion of the first phase, each participant will take a probiotic mixture containing Bifidobacterium longum Rosell®-175 & Lactobacillus helveticus Rosell®-52 and excipients: potato starch, magnesium stearate, and the capsule shell of hydroxypropyl methylcellulose. (Sanprobi Stress; Sanprobi sp. z o.o., sp.k., Szczecin, Poland) for another 3 months.
  * Dosage: One capsule per day, containing 3 × 10⁹ (3 billion) CFU*.
  * Instructions: Take before 1:00 PM. Do not consume hot drinks immediately after taking the capsule.
  * CFU = Colony Forming Units
  Arms: Anti-inflammatory diet + placebo first; Pro-inflammatory diet + placebo first

SUMMARY:
The goal of this study is to explore the potential impact of an anti-inflammatory probiotic mixture of psychobiotics including Bifidobacterium longum Rosell®-175 and Lactobacillus helveticus Rosell®-52 on cognitive functions in older adults following either pro-inflammatory or anti-inflammatory diets. According to recent findings, even short-term exposure to foods with pro- or anti-inflammatory properties may lead to corresponding negative or beneficial effects on cognitive functioning .

The main questions this study aims to answer are:

* How important is the initial dietary pattern for observing possible beneficial effects of probiotic supplementation? (Diet as a potential moderator)
* How important is the initial state of the gut microbiota for observing possible beneficial effects of probiotic supplementation? (Microbiota as a potential moderator)
* Is it possible to improve or slow down the decline in cognitive functions associated with aging with probiotic supplementation?
* Can probiotic supplementation counteract the negative effects of pro-inflammatory dietary patterns?

The investigators will compare probiotic to a placebo (a look-alike substance that contains no active ingredients) to determine whether probiotic is effective in enhancing cognitive function.

Participants:

* Take a probiotic or placebo capsule daily for 3 months
* Undergo a crossover after 3 months - those who initially took probiotics will switch to the placebo, and vice versa
* Visit SWPS University for screening (T0), baseline assessments before beginning supplementation (T1), and follow-up assessments at 3 months (T2) and 6 months (T3). The T2 visit occurs just before the crossover.
* Complete neuropsychological testing, questionnaires, and EEG recordings during the T1, T2, and T3 visits.
* Provide stool samples for gut microbiota analysis at the T1, T2, and T3 visits.
* Maintain their usual dietary habits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or older
* Signed written Informed Consent Form
* Score ≥28 on the Mini-Mental State Examination (MMSE)
* A willingness and motivation to follow the study protocol

Exclusion Criteria:

* Regular use of prebiotics, antibiotics, or antifungal medications
* Use of prebiotics, antibiotics, or antifungal medications within the past 3 months
* Diagnosed neurological disorder
* History of head injury with neurological consequences
* Left-handedness

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Differentiation score in California Verbal Learning Test (CVLT) to assess long-term memory | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  California Verbal Learning Test (CVLT) measure the verbal learning and memory. It measures how well individuals learn and recall verbal material, assessing both short-term and long-term memory. The Differentiation score measures the ability to distinguish between correct and incorrect responses. Scores range from 0 to 16, with higher scores indicating better outcome.
Change in d' score in old/new recognition test (ONR) to assess long-term memory | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  The old/new word recognition task is designed to assess episodic memory. It is consisted of two phases: a learning phase and a recognition phase. During the learning phase, participants viewed 30 pictures on the computer. In the recognition phase, participants were presented with 30 "old" and 30 "new" pictures in random order and were asked to determine whether each picture had been shown during the learning phase.
  To analyze episodic memory task we followed Macmillan and Creelman (2005) signal detection theory, where d' is the ability to discriminate between signal and noise (between old and new stimuli), H stands for the proportion of correct changes detected (hit rate), and F stands for the proportion of changes incorrectly reported (false alarm rate).
  d' = zH - zF
Change in N400 event-related potential (ERP) component amplitude to assess long-term memory | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  The N400 ERP component will be measured during an old/new word recognition task designed to assess episodic memory. The task involves presenting participants with previously studied ("old") and novel ("new") words while EEG is recorded. The N400 component-typically observed as a negative deflection peaking around 400 ms post-stimulus-is sensitive to familiarity and memory retrieval. A reduced N400 amplitude for old versus new words is interpreted as successful recognition. Changes in N400 amplitude over time will indicate modulation of episodic memory performance across the intervention.

SECONDARY OUTCOMES:
Changes in Beck Depression Inventory (BDI) total score to assess symptoms of depression | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Changes in the Fatigue Assessment Scale (FAS) total score to assess symptoms of chronic fatigue | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 10 to 50, with higher scores indicating greater fatigue.
Change in the number of correctly marked target characters in the d2 Test of Attention (d2-R) - to assess attention. | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 308, with higher scores indicating better outcome.
Change in Concentration score in d2 Test of Attention (d2-R) - to assess attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 308, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Symbol Substitution subtest total score to assess cognitive processing speed, visual-motor coordination, and sustained attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 39, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Span Forward subset total score to assess short-term auditory memory | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 14, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Span Backward subset total score to assess short-term auditory memory | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 14, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Block Design subtest total score to assess visual domains such as visuoperceptive, visuospatial and visuoconstructive functions | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  Scores range from 0 to 54, with higher scores indicating better outcome.
Change in Color Trails Test (CTT) total mistakes - CTT1 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  There is no predefined maximum number of errors in the test.
Change in Color Trails Test (CTT) total mistakes - CTT2 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  There is no predefined maximum number of errors in the test.
Change in Color Trails Test (CTT) completion time - CTT1 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  A maximum time limit of 240 seconds (4 minutes) is applied.
Change in Color Trails Test (CTT) completion time - CTT2 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
  A maximum time limit of 240 seconds (4 minutes) is applied.
Change in Color Trails Test (CTT) Interference score - to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
Change in P300 event-related potential (ERP) component amplitude to assess attention | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
Changes in diversity in microbial community in a single sample (alpha-diversity) | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
Changes in diversity in microbial community between samples (beta-diversity) | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.
Changes in differential abundance of microbial community | Baseline (prior to intervention), at the end of the 3-month probiotic/placebo supplementation period, and again 3 months after the crossover.

OTHER OUTCOMES:
Dietary inflammatory index | Baseline (prior to intervention)
  Dietary Inflammatory Index assessment based on the Shivappa et al. (2014) equation. It classifies participants' dietary patterns as pro-inflammatory, neutral, or anti-inflammatory. Scores ranged from -8.87 (maximally anti-inflammatory diet) to +7.98 (maximally pro-inflammatory diet).
Score in Mini-mental state examination (MMSE) | Baseline (prior to intervention)
  A screening tool for cognitive impairment with older adults. It is scored on a scale from 0 to 30.
  27-30 points: Normal result, no cognitive impairment 24-26 points: Cognitive impairment without dementia 19-23 points: Mild dementia 11-18 points: Moderate dementia 0-10 points: Severe dementia
Score in the Raven's Progressive Matrices test | Baseline (prior to intervention)
  The Raven's Progressive Matrices test is used to measure the level of general intelligence, understood as fluid intelligence. It is scored on a scale from 0 to 60, with higher scores indicating better outcome.
Score in Adherence to the Mediterranean diet | Baseline (prior to intervention)
  The scale ranges from 0 to 7, with higher scores reflecting greater adherence to the Mediterranean diet.

CONTACTS AND LOCATIONS:
Locations (1):
- SWPS University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes